CLINICAL TRIAL: NCT02600546
Title: Evaluation of the Repeatability and Reproducibility of Corneal Epithelial Thickness Mapping With SD-OCT
Status: Completed | Type: Observational
Sponsor: Optovue (Industry)
Responsible Party: Sponsor
Other Study IDs: 200-50545
Record Dates: First submitted 2015-11-05; First posted 2015-11-09 (Estimated); Last update posted 2016-03-30 (Estimated); Status verified 2015-11

CONDITIONS: Repeatability & Reproducibility

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Prospective

SUMMARY:
Evaluate the repeatability and reproducibility of the RTVue-XR for measuring the total corneal thickness (pachymetry), the epithelial thickness, and the stromal thickness mapping in normal subjects and corneal patients.

ELIGIBILITY:
Inclusion Criteria:

* Able and willing to provide consent.
* Able and willing to complete required exams
* History of refractive surgery, contact lens, dry eye or keratoconus for corneal patients

Exclusion Criteria:

* Unable to complete required exams
* History of refractive surgery, contact lens, dry eye or keratoconus for normal patients

Min Age: 18 Years | Sex: All | Healthy Volunteers: Yes
Age Groups: Adult, Older Adult
Study Population: Seeing eye doctor for routine or follow-up care
Sampling Method: Non-Probability Sample
Enrollment: 62 (Actual)
Dates: Start 2015-10; Primary Completion 2016-02 (Actual); Study Completion 2016-02 (Actual)

PRIMARY OUTCOMES:
epithelial thickness | Day 1

SECONDARY OUTCOMES:
Stromal thickness | Day 1

CONTACTS AND LOCATIONS:
Locations (1):
- Baylor College of Medicine, Houston, Texas, United States